CLINICAL TRIAL: NCT02217410
Title: A 12-month Randomized, Multiple Dose, Open-label, Study Evaluating Safety, Tolerability, Pharmacokinetics/Pharmacodynamics (PK/PD) and Efficacy of an Anti-CD40 Monoclonal Antibody, CFZ533, in Combination With Mycophenolate Mofetil (MMF) and Corticosteroids (CS), With and Without Tacrolimus (Tac), in de Novo Renal Transplant Recipients
Brief Title: CCFZ533X2201 - PoC Study in de Novo Renal Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CCFZ533X2201
Record Dates: First submitted 2014-08-07; First posted 2014-08-15 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Kidney Transplantation
Keywords: renal, de novo,
MeSH Terms: interventions — iscalimab; Tacrolimus; Triamcinolone; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Regimen A (Experimental): CFZ533 administered with the contemporary standard of care (SoC) consists of concentration-controlled tacrolimus (Tac), combined with mycophenolate mofetil (MMF) and corticosteroids (CS).
  Interventions: Biological: CFZ533; Drug: Tacrolimus (Tac); Drug: Mycophenolate mofetil (MMF); Drug: Corticosteroids (CS)
- Regimen B (Experimental): CFZ533 administered with mycophenolate mofetil (MMF) and corticosteroids (CS) with anti-IL2 induction
  Interventions: Biological: CFZ533; Drug: Mycophenolate mofetil (MMF); Drug: Corticosteroids (CS); Biological: anti-IL2 Induction
- Regimen C (Active Comparator): Standard of care (SoC) [concentration-controlled tacrolimus (Tac) combined with mycophenolate mofetil (MMF) and corticosteroids (CS) with anti-IL2 induction]
  Interventions: Drug: Tacrolimus (Tac); Drug: Mycophenolate mofetil (MMF); Drug: Corticosteroids (CS); Biological: anti-IL2 Induction

INTERVENTIONS:
Biological: CFZ533
  Arms: Regimen A; Regimen B
Drug: Tacrolimus (Tac)
  Arms: Regimen A; Regimen C
Drug: Mycophenolate mofetil (MMF)
Drug: Corticosteroids (CS)
Biological: anti-IL2 Induction
  Arms: Regimen B; Regimen C

SUMMARY:
The purpose of this study was to investigate the safety, tolerability, pharmacokinetics (PK) and potential for CFZ533 to replace calcineurin inhibitors (CNI), while providing a similar rate of acute rejection prophylaxis and renal function in a de novo renal transplant population receiving an allograft from standard criteria donors.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Recipients of a kidney transplant from a heart-beating deceased, living unrelated or non-human leukocyte antigen (HLA) identical living related donor.
* Recipients of a kidney with a cold ischemia time (CIT) < 30 hours.

Main Exclusion Criteria:

* Recipients of an organ from a non-heart beating donor.
* ABO incompatible or complement-dependent lymphocytotoxic (CDC) crossmatch positive transplant.
* Subjects receiving a second kidney allograft, unless the first allograft was lost due to surgical complication.
* Subjects at high immunological risk for rejection
* Subjects at risk for tuberculosis (TB)
* Subject with severe systemic infections, current or within the two weeks prior to randomization/enrollment.
* Any additional contraindication to the use of tacrolimus or mycophenolate mofetil according to the national labeling information of these products (see local product label).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (6):
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Livingston, New Jersey
  - Novartis Investigative Site, Cincinnati, Ohio
- Novartis Investigative Site, São Paulo, São Paulo, Brazil
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
- Netherlands (3):
  - Novartis Investigative Site, Utrecht, The Netherlands
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=420

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Part 1, patients were enrolled into Arm 1. In Part 2, patients were randomized (2:1) to Arms 2A and 2B.
Pre-assignment Details: Study Part 1 focused on measuring the multiple-dose safety, tolerability, PK, and PD of both IV and SC CFZ533 when administered with the SoC treatment regimen.
  Study Part 2 investigated efficacy, safety, tolerability, PK and PD of CFZ533 in the absence of Tac.
Groups:
- CFZ533 + TAC + MMF (Part 1): CFZ533 (3 mg/kg SC) administered with the contemporary standard of care (SoC) consists of concentration-controlled tacrolimus (Tac), combined with mycophenolate mofetil (MMF) and corticosteroids (CS).
- CFZ533 + MMF (Part 2): CFZ533 (10mg/kg IV) administered with mycophenolate mofetil (MMF) and corticosteroids (CS) with anti-IL2 induction
- Tac + MMF (Part 2): Standard of care (SoC) [concentration-controlled tacrolimus (Tac) combined with mycophenolate mofetil (MMF) and corticosteroids (CS) with anti-IL2 induction]
Period: Overall Study
Arm/Group | CFZ533 + TAC + MMF (Part 1) | CFZ533 + MMF (Part 2) | Tac + MMF (Part 2)
Started | 7 | 34 | 18
Completed | 6 | 30 | 13
Not Completed | 1 | 4 | 5
Not completed — Graft Loss | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Physician Decision | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all patients that received at least one dose of study drug.
  For Part 2, all patients that received their transplant along with any patient who received study drug but had no transplant were combined.
Groups:
- Total: Total of all reporting groups
Arm/Group | CFZ533 + TAC + MMF (Part 1) | CFZ533 + MMF (Part 2) | Tac + MMF (Part 2) | Total
Number analyzed (Participants) | 7 | 34 | 18 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (9.30) | 49.0 (15.79) | 53.4 (18.01) | 50.1 (15.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 6 | 17
  Male | 4 | 26 | 12 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 20 | 9 | 31
  Unknown or Not Reported | 5 | 13 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Mean Cmax Pharmacokinetic Parameter- Part I
Description: Pharmacokinetics as defined by the systemic concentrations and Cmax of certain immunosuppressant medications used in Part I
Time Frame: Day 1
Population: The PK Analysis Set included all patients with at least one available valid (i.e., not flagged for exclusion) PK concentration measurement, who received study drug and experienced no protocol deviations with relevant impact on PK data.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | CFZ533 + TAC + MMF (Part 1)
Number analyzed (Participants) | 7
ug/mL | 66.3 (12.3)

2. Primary Outcome: Mean Tmax Pharmacokinetic Parameter - Part I
Description: Quantify pharmacokinetics of CFZ533 in combination with MMF, CS, and tacrolimus in de novo renal transplant patients during the treatment and follow-up periods.
Time Frame: Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: day
Arm/Group | CFZ533 + TAC + MMF (Part 1)
Number analyzed (Participants) | 7
day | 0.237 [0 to 1.02]

3. Primary Outcome: Mean AUClast Pharmacokinetic Parameter - Part I
Description: as for outcome 2
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | CFZ533 + TAC + MMF (Part 1)
Number analyzed (Participants) | 7
day*ug/mL | 367 (52.0)

4. Primary Outcome: Efficacy as Defined by the Frequency and Severity (Banff Classification) of Treated Biopsy Proven Acute Rejection (tBPAR) Adjudicated Data - Part II
Description: To assess the activity of the investigational arm as compared to the standard of care control arm in de novo renal transplant patients as measured by the frequency and severity of tBPAR as measured on the Banff classification scale.
  An adjudication was performed on all on cause renal biopsies by an independent expert committee blinded to therapy.
Time Frame: 3, 6, 9, and 12 months
Population: PD analysis set included all Patients in the Full Analysis set with available PD data and no protocol deviations with relevant impact on PD data.
Measure: Number; unit: events
Arm/Group | CFZ533 + MMF (Part 2) | Tac + MMF (Part 2)
Number analyzed (Participants) | 33 | 18
events
  Month 3 | 6 | 2
  Month 6 | 7 | 3
  Month 9 | 7 | 3
  Month 12 | 7 | 3
Statistical Analysis 1: Comparison: CFZ533 + MMF (Part 2) vs Tac + MMF (Part 2); Test type: Other; p = 0.8976, Bayesian posterior probability; Posterior probability that the composite efficacy failure difference between CFZ533 and Tac is < 20%; Mean Difference (Final Values) = 0.095, 95% CI 2-sided [-0.067 to 0.263] — Month 3
Statistical Analysis 2: Comparison: CFZ533 + MMF (Part 2) vs Tac + MMF (Part 2); Test type: Other; p = 0.8836, Bayesian posterior probability; Posterior probability that the composite efficacy failure difference between CFZ533 and Tac is < 20%; Mean Difference (Final Values) = 0.093, 95% CI 2-sided [-0.084 to 0.271] — Month 6
Statistical Analysis 3: Comparison: CFZ533 + MMF (Part 2) vs Tac + MMF (Part 2); Test type: Other; p = 0.8822, Bayesian posterior probability; Posterior probability that the composite efficacy failure difference between CFZ533 and Tac is < 20%; Mean Difference (Final Values) = 0.093, 95% CI 2-sided [-0.085 to 0.272] — Month 9
Statistical Analysis 4: Comparison: CFZ533 + MMF (Part 2) vs Tac + MMF (Part 2); Test type: Other; p = 0.8821, Bayesian posterior probability; Posterior probability that the composite efficacy failure difference between CFZ533 and Tac is < 20%; Mean Difference (Final Values) = 0.093, 95% CI 2-sided [-0.087 to 0.273] — Month 12

5. Secondary Outcome: Total Soluble CD40 and Total Soluble CD154 Concentrations in Plasma - Part 1
Description: To quantify the change from baseline and recovery of peripheral blood total soluble CD40 and total soluble CD154
Time Frame: Baseline to end of study (Day 1, Day 29, Day 337)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- sCD40 (Part I); sCD154: CFZ533 (3 mg/kg SC) administered with the contemporary standard of care (SoC) consists of concentration-controlled tacrolimus (Tac), combined with mycophenolate mofetil (MMF) and corticosteroids (CS).
Arm/Group | sCD40 (Part I) | sCD154
Number analyzed (Participants) | 7 | 7
ng/ml
  Baseline: number analyzed (Participants) | 3 | 3
  Baseline | 4.03 (4.08) | 0.125 (0.007)
  Day 1: number analyzed (Participants) | 6 | 6
  Day 1 | 8.86 (0.0585) | 0.0585 (0.0711)
  Day 2 | 16.7 (4.51) | 0.139 (0.193)
  Day 3 | 24.8 (4.47) | 0.157 (0.235)
  Day 4 | 31.3 (6.34) | 0.241 (0.418)
  Day 8 | 54.0 (11.2) | 0.399 (0.636)
  Day 15 | 84.1 (13.8) | 0.0879 (0.139)
  Day 22 | 102 (13.9) | 0.0500 (0.132)
  Day 29: number analyzed (Participants) | 7 | 6
  Day 29 | 120 (15.7) | 0.225 (0.504)
  Day 36 | 128 (19.2) | 0.116 (0.2)
  Day 43: number analyzed (Participants) | 6 | 6
  Day 43 | 145 (25.6) | 0.0193 (0.0474)
  Day 50: number analyzed (Participants) | 5 | 5
  Day 50 | 156 (6.35) | 0.0478 (0.0687)
  Day 57: number analyzed (Participants) | 6 | 5
  Day 57 | 161 (21.2) | 0 (0)
  Day 64: number analyzed (Participants) | 6 | 6
  Day 64 | 163 (24.2) | 0.0316 (0.0492)
  Day 71: number analyzed (Participants) | 6 | 6
  Day 71 | 156 (19.2) | 0.0148 (0.0363)
  Day 85: number analyzed (Participants) | 6 | 6
  Day 85 | 168 (21.4) | 0.0139 (0.0340)
  Day 99: number analyzed (Participants) | 6 | 6
  Day 99 | 155 (23.3) | 0 (0)
  Day 113: number analyzed (Participants) | 6 | 6
  Day 113 | 85.7 (47.9) | 0.0668 (0.164)
  Day 127: number analyzed (Participants) | 6 | 5
  Day 127 | 12.2 (15.7) | 0.0488 (0.0697)
  EoS: number analyzed (Participants) | 6 | 5
  EoS | 0.918 (0.330) | 0.0184 (0.0411)

6. Secondary Outcome: Free CD40 and Total CD40 on B Cells - Part II
Description: The magnitude and duration of peripheral blood CD40 occupancy. MESF: molecules of equivalent soluble fluorochrome
Time Frame: Baseline to end of study (Day 1/predose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: MESF
Groups:
- Free CD40 on Whole Blood B Ceels; Total CD40 on Whole Blood B Cells: CFZ533 (10mg/kg IV) administered with mycophenolate mofetil (MMF) and corticosteroids (CS) with anti-IL2 induction
Arm/Group | Free CD40 on Whole Blood B Ceels | Total CD40 on Whole Blood B Cells
Number analyzed (Participants) | 26 | 29
MESF
  CFZ553 + MMF (Baseline): number analyzed (Participants) | 25 | 25
  CFZ553 + MMF (Baseline) | 30836.00 (13648.69) | 12778.80 (7873.76)
  CFZ553 + MMF (D1 - 6h post dose) | 1623.81 (1359.85) | 13806.90 (7185.66)
  CFZ553 + MMF (D15): number analyzed (Participants) | 22 | 26
  CFZ553 + MMF (D15) | 799.62 (762.38) | 15160.38 (7398.57)
  CFZ553 + MMF (D 29): number analyzed (Participants) | 19 | 25
  CFZ553 + MMF (D 29) | 817.63 (1540.16) | 13299.60 (6330.89)
  CFZ553 + MMF (D 57): number analyzed (Participants) | 22 | 24
  CFZ553 + MMF (D 57) | 597.13 (523.55) | 12234.38 (6943.13)
  CFZ553 + MMF (D 85): number analyzed (Participants) | 19 | 22
  CFZ553 + MMF (D 85) | 635.47 (614.68) | 9330.86 (8484.46)
  CFZ553 + MMF (D 197): number analyzed (Participants) | 12 | 14
  CFZ553 + MMF (D 197) | 3699.0 (7298.98) | 2820.72 (2347.11)
  CFZ553 + MMF (253): number analyzed (Participants) | 16 | 7
  CFZ553 + MMF (253) | 2667.38 (6146.86) | 1427.14 (740.48)
  CFZ553 + MMF (EoS): number analyzed (Participants) | 18 | 12
  CFZ553 + MMF (EoS) | 176.17 (266.82) | 1069.67 (809.12)
  Tac + MMF (Baseline): number analyzed (Participants) | 12 | 14
  Tac + MMF (Baseline) | 31508.33 (12759.49) | 14581.43 (9342.79)
  Tac + MMF (D1 - 6h post dose): number analyzed (Participants) | 17 | 16
  Tac + MMF (D1 - 6h post dose) | 26437.65 (11930.50) | 13715.00 (8293.33)
  Tac + MMF (D15): number analyzed (Participants) | 12 | 14
  Tac + MMF (D15) | 24441.67 (9125.93) | 13707.14 (6770.14)
  Tac + MMF (D29): number analyzed (Participants) | 15 | 16
  Tac + MMF (D29) | 27840.00 (12106.72) | 12698.75 (6002.96)
  Tac + MMF (D57): number analyzed (Participants) | 14 | 13
  Tac + MMF (D57) | 27994.29 (12004.57) | 12583.85 (6210.07)
  Tac + MMF (D85): number analyzed (Participants) | 15 | 13
  Tac + MMF (D85) | 25044.00 (10896.65) | 8701.54 (4183.00)
  Tac + MMF (D197): number analyzed (Participants) | 10 | 5
  Tac + MMF (D197) | 21360.00 (3155.67) | 2067.60 (1617.28)
  Tac + MMF (D253): number analyzed (Participants) | 8 | 8
  Tac + MMF (D253) | 15752.75 (7145.32) | 1750.50 (1005.84)
  Tac + MMF (EoS): number analyzed (Participants) | 9 | 6
  Tac + MMF (EoS) | 21200.00 (4407.95) | 6276.17 (11271.20)

7. Secondary Outcome: Anti-CFZ533 Antibodies - Part I
Description: To evaluate the immunogenicity of CFZ533 via the quantitative analysis of anti-CFZ533 antibodies
Time Frame: Baseline to end of study
Population: Safety analysis set included all patients that received at least one dose of study drug.
Measure: Number; unit: anti-CFZ533 antibodies
Arm/Group | CFZ533 + TAC + MMF (Part 1)
Number analyzed (Participants) | 7
anti-CFZ533 antibodies | 0

8. Secondary Outcome: Anti-CFZ533 Antibodies - Part II
Description: To evaluate the immunogenicity of CFZ533 via the quantitative analysis of anti-CFZ533 antibodies
Time Frame: Baseline to end of study (screening, baseline, Day 141, Day 225, Day 309, Study Completion)
Population: Safety analysis set included all patients that received at least one dose of study drug. For Part 2, all patients that received their transplant along with any patient who received study drug but had no transplant were combined.
Measure: Number; unit: anti-CFZ533 antibodies
Arm/Group | CFZ533 + MMF (Part 2) | Tac + MMF (Part 2)
Number analyzed (Participants) | 34 | 18
anti-CFZ533 antibodies
  Screening: number analyzed (Participants) | 31 | 16
  Screening | 0 | 0
  Baseline: number analyzed (Participants) | 6 | 0
  Baseline | 0 |
  Day 141: number analyzed (Participants) | 22 | 11
  Day 141 | 0 | 0
  Day 225: number analyzed (Participants) | 21 | 10
  Day 225 | 0 | 0
  Day 309: number analyzed (Participants) | 20 | 8
  Day 309 | 0 | 0
  Study Completion: number analyzed (Participants) | 21 | 10
  Study Completion | 0 | 0

9. Secondary Outcome: eGFR - Part II
Description: Renal function as assessed by MDRD (Modification of Diet in Renal Disease) formula.
  eGFR: Estimated glomerular filtration rate
Time Frame: Day 1, Day 29, Day 337,
Population: as for outcome 8
Measure: Mean (90% Confidence Interval); unit: ml/min
Arm/Group | CFZ533 + MMF (Part 2) | Tac + MMF (Part 2)
Number analyzed (Participants) | 32 | 18
ml/min
  Day 1 | 9.8 [8.3 to 11.3] | 9.7 [7.7 to 11.8]
  Day 29: number analyzed (Participants) | 30 | 16
  Day 29 | 55.6 [50.4 to 60.7] | 44.3 [37.2 to 51.4]
  Day 337: number analyzed (Participants) | 20 | 10
  Day 337 | 58.2 [52.2 to 64.2] | 44.2 [36.1 to 52.3]

10. Secondary Outcome: CFZ533 Plasma PK Concentrations - Part II
Description: Quantify the systemic concentrations of CFZ533 in combination with MMF, CS, and tacrolimus in de novo renal transplant patients during the treatment and follow-up periods. A full pharmacokinetic analysis can be performed on the concentration-time data to evaluate the impact of renal transplantation on the various medications used in the treatment regimen.
Time Frame: throughout study period (day 84 to day 336)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | CFZ533 + MMF (Part 2)
Number analyzed (Participants) | 32
ug/mL
  Day 84: number analyzed (Participants) | 23
  Day 84 | 247 (58.2)
  Day 112: number analyzed (Participants) | 24
  Day 112 | 211 (51.8)
  Day 140: number analyzed (Participants) | 23
  Day 140 | 178 (54.9)
  Day 168: number analyzed (Participants) | 23
  Day 168 | 157 (57.4)
  Day 196: number analyzed (Participants) | 23
  Day 196 | 148 (53.1)
  Day 224: number analyzed (Participants) | 21
  Day 224 | 147 (53.8)
  Day 252: number analyzed (Participants) | 22
  Day 252 | 151 (35.2)
  Day 280: number analyzed (Participants) | 22
  Day 280 | 160 (87.7)
  Day 308: number analyzed (Participants) | 22
  Day 308 | 132 (42.5)
  Day 336: number analyzed (Participants) | 21
  Day 336 | 156 (85.2)
  End of study: number analyzed (Participants) | 21
  End of study | 133 (57.8)

11. Secondary Outcome: Total sCD40 Plasma Concentrations - Part II
Description: To quantify the change from baseline and recovery of peripheral blood total soluble CD40
Time Frame: 12 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CFZ533 + MMF (Part 2) | Tac + MMF (Part 2)
Number analyzed (Participants) | 32 | 17
ng/mL
  Baseline: number analyzed (Participants) | 30 | 15
  Baseline | 3.02 (2.44) | 3.67 (2.15)
  Day 1: number analyzed (Participants) | 32 | 15
  Day 1 | 6.95 (4.29) | 1.16 (1.15)
  Day 4: number analyzed (Participants) | 31 | 17
  Day 4 | 24.6 (11.0) | 1.16 (1.15)
  Day 15: number analyzed (Participants) | 31 | 17
  Day 15 | 69.6 (21.5) | 0.869 (1.55)
  Day 29: number analyzed (Participants) | 31 | 15
  Day 29 | 101 (18.9) | 0.362 (0.0746)
  Day 57: number analyzed (Participants) | 26 | 15
  Day 57 | 140 (17.4) | 0.438 (0.316)
  Day 85: number analyzed (Participants) | 24 | 16
  Day 85 | 189 (76.4) | 0.429 (0.324)
  Day 113: number analyzed (Participants) | 24 | 15
  Day 113 | 215 (75.5) | 0.391 (0.129)
  Day 141: number analyzed (Participants) | 22 | 15
  Day 141 | 237 (93.1) | 0.453 (0.271)
  Day 169: number analyzed (Participants) | 23 | 15
  Day 169 | 238 (80.3) | 0.537 (0.215)
  Day 197: number analyzed (Participants) | 22 | 12
  Day 197 | 253 (81.3) | 0.423 (0.0908)
  Day 225: number analyzed (Participants) | 19 | 12
  Day 225 | 258 (77.7) | 0.452 (0.119)
  Day 253: number analyzed (Participants) | 20 | 11
  Day 253 | 236 (36.5) | 0.457 (0.0800)
  Day 281: number analyzed (Participants) | 21 | 12
  Day 281 | 273 (71.3) | 0.455 (0.0789)
  Day 309: number analyzed (Participants) | 22 | 11
  Day 309 | 286 (66.0) | 0.454 (0.0957)
  Day 337: number analyzed (Participants) | 22 | 11
  Day 337 | 298 (57.4) | 0.411 (0.0581)
  End of Study: number analyzed (Participants) | 20 | 12
  End of Study | 303 (59.7) | 0.959 (1.88)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 3 years.
Groups:
- Total: Total
Arm/Group | CFZ533 + TAC + MMF (Part 1) | CFZ533 + MMF (Part 2) | Tac + MMF (Part 2) | Total
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/34 | 0/18 | 0/59
Serious Adverse Events (participants affected / at risk) | 4/7 | 21/34 | 12/18 | 37/59
Other Adverse Events (participants affected / at risk) | 7/7 | 33/34 | 18/18 | 58/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CFZ533 + TAC + MMF (Part 1) (N=7) | CFZ533 + MMF (Part 2) (N=34) | Tac + MMF (Part 2) (N=18) | Total (N=59)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 1
Photophobia (Eye disorders) | 1 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 3
Kidney transplant rejection (Immune system disorders) | 0 | 5 | 1 | 6
Transplant rejection (Immune system disorders) | 0 | 2 | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 3 | 2 | 5
Encephalitis (Infections and infestations) | 0 | 0 | 1 | 1
Enterobacter bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 1
Hepatitis C (Infections and infestations) | 0 | 1 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Polyomavirus-associated nephropathy (Infections and infestations) | 0 | 4 | 1 | 5
Pyelonephritis (Infections and infestations) | 0 | 2 | 3 | 5
Renal cyst infection (Infections and infestations) | 0 | 1 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 2 | 2
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 4
Delayed graft function (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Graft loss (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Transplant failure (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Amylase increased (Investigations) | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 2
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 2
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 1
Lymphocele (Vascular disorders) | 0 | 0 | 1 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CFZ533 + TAC + MMF (Part 1) (N=7) | CFZ533 + MMF (Part 2) (N=34) | Tac + MMF (Part 2) (N=18) | Total (N=59)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 4 | 8
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 3 | 2 | 6
Leukopenia (Blood and lymphatic system disorders) | 1 | 13 | 3 | 17
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 3
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 1 | 2
Arrhythmia (Cardiac disorders) | 0 | 2 | 1 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 1 | 3
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 4 | 1 | 7
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 2 | 0 | 1 | 3
Chalazion (Eye disorders) | 0 | 1 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 0 | 1
Eye movement disorder (Eye disorders) | 2 | 0 | 0 | 2
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 3 | 7
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 5 | 0 | 5
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 14 | 8 | 23
Diarrhoea (Gastrointestinal disorders) | 2 | 8 | 10 | 20
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 1 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gingival recession (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 10 | 9 | 23
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Paraesthesia oral (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Tongue discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 8 | 4 | 15
Asthenia (General disorders) | 0 | 0 | 1 | 1
Catheter site pain (General disorders) | 0 | 0 | 2 | 2
Chills (General disorders) | 0 | 3 | 0 | 3
Cyst (General disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 5 | 5 | 11
Generalised oedema (General disorders) | 1 | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 2 | 1 | 3
Influenza like illness (General disorders) | 1 | 0 | 0 | 1
Infusion site swelling (General disorders) | 0 | 1 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 2 | 7 | 6 | 15
Pain (General disorders) | 1 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 2
Secretion discharge (General disorders) | 3 | 0 | 0 | 3
Swelling (General disorders) | 0 | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 1
Kidney transplant rejection (Immune system disorders) | 0 | 0 | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
BK virus infection (Infections and infestations) | 3 | 10 | 6 | 19
Bronchitis (Infections and infestations) | 0 | 4 | 0 | 4
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 6 | 2 | 8
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 2 | 2
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 2
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 1 | 2
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 2
Human polyomavirus infection (Infections and infestations) | 0 | 2 | 0 | 2
Infection (Infections and infestations) | 0 | 1 | 1 | 2
Influenza (Infections and infestations) | 0 | 2 | 1 | 3
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 1
Latent tuberculosis (Infections and infestations) | 0 | 0 | 1 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1 | 1
Mucocutaneous candidiasis (Infections and infestations) | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 10 | 4 | 15
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1
Oral infection (Infections and infestations) | 0 | 1 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 2
Polyomavirus-associated nephropathy (Infections and infestations) | 0 | 3 | 1 | 4
Pyelonephritis (Infections and infestations) | 0 | 1 | 1 | 2
Pyuria (Infections and infestations) | 0 | 1 | 1 | 2
Respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 1 | 2
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 0 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 8 | 7 | 16
Urinary tract infection viral (Infections and infestations) | 0 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 1
Wound infection bacterial (Infections and infestations) | 0 | 1 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 | 3 | 2 | 5
Delayed graft function (Injury, poisoning and procedural complications) | 0 | 3 | 3 | 6
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Graft complication (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Incision site complication (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Incision site erythema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Incision site pain (Injury, poisoning and procedural complications) | 3 | 6 | 2 | 11
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 5 | 1 | 6
Procedural pain (Injury, poisoning and procedural complications) | 0 | 3 | 6 | 9
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 | 2 | 3 | 5
Wound complication (Injury, poisoning and procedural complications) | 0 | 11 | 8 | 19
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Wound haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Amylase increased (Investigations) | 0 | 3 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 2
Blood creatinine increased (Investigations) | 0 | 3 | 1 | 4
Blood glucose increased (Investigations) | 0 | 1 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 1
Blood phosphorus decreased (Investigations) | 1 | 0 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 1 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 1
Cardiac murmur (Investigations) | 1 | 0 | 0 | 1
Cytomegalovirus test positive (Investigations) | 0 | 1 | 0 | 1
Drug level decreased (Investigations) | 0 | 0 | 1 | 1
Electrocardiogram ST segment abnormal (Investigations) | 1 | 0 | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 1 | 3
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 1
Heart rate irregular (Investigations) | 0 | 1 | 0 | 1
Lipase increased (Investigations) | 0 | 2 | 0 | 2
Polyomavirus test positive (Investigations) | 0 | 1 | 0 | 1
Vitamin D decreased (Investigations) | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 1 | 1 | 0 | 2
Weight increased (Investigations) | 0 | 2 | 1 | 3
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 1
White blood cell count increased (Investigations) | 0 | 3 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4 | 1 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 3 | 3 | 6
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4 | 4 | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 9 | 5 | 15
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 4
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 5
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 6 | 5 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 3 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 11 | 5 | 21
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 2 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 2 | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 1 | 6
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 5
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 6 | 1 | 8
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 3 | 6
Dizziness postural (Nervous system disorders) | 1 | 0 | 1 | 2
Headache (Nervous system disorders) | 1 | 6 | 4 | 11
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 2
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 2 | 3 | 6 | 11
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 2
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 11 | 5 | 17
Mood swings (Psychiatric disorders) | 0 | 1 | 0 | 1
Phonophobia (Psychiatric disorders) | 1 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 1
Bladder pain (Renal and urinary disorders) | 0 | 0 | 1 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 3 | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 2 | 3
Leukocyturia (Renal and urinary disorders) | 0 | 1 | 1 | 2
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 1 | 0 | 2
Perinephric collection (Renal and urinary disorders) | 0 | 2 | 0 | 2
Perinephric oedema (Renal and urinary disorders) | 0 | 0 | 1 | 1
Polyuria (Renal and urinary disorders) | 0 | 5 | 0 | 5
Proteinuria (Renal and urinary disorders) | 0 | 2 | 1 | 3
Renal impairment (Renal and urinary disorders) | 0 | 0 | 2 | 2
Renal tubular acidosis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal tubular injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 2 | 2
Sterile pyuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urethral pain (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 2 | 3
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary tract disorder (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 2 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Penile oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 10 | 2 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 5
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 3
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3
Pityriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 2 | 0 | 2
Hot flush (Vascular disorders) | 0 | 2 | 0 | 2
Hypertension (Vascular disorders) | 1 | 13 | 6 | 20
Hypotension (Vascular disorders) | 0 | 2 | 3 | 5
Lymphocele (Vascular disorders) | 0 | 1 | 1 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 1
Poor venous access (Vascular disorders) | 0 | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT02217410/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT02217410/SAP_001.pdf